CLINICAL TRIAL: NCT06358937
Title: Clinical and Microbiological Evaluation of Laser Assisted New Attachment Procedure (LANAP) Using Nd:Yag vs. Diode Laser in the Management Of Stage II Periodontitis (Randomized Controlled Clinical Trial)
Brief Title: Clinical and Microbiological Evaluation of Laser Assisted New Attachment Procedure (LANAP) Using Nd:Yag vs. Diode Laser in the Management Of Stage II Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Salem (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Salem, Master's candidate of Periodontology, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #7/2023
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Assisted New Attachment Procedure using ND:YAG laser (Experimental)
  Interventions: Device: Laser Assisted New Attachment Procedure using ND:YAG laser
- Laser Assisted New Attachment Procedure using diode laser (Experimental)
  Interventions: Device: Laser Assisted New Attachment Procedure using diode laser
- Scaling and Root Planing using ultrasonic and curettes (Active Comparator)
  Interventions: Procedure: Scaling and Root Planing using ultrasonic and curettes

INTERVENTIONS:
Device: Laser Assisted New Attachment Procedure using ND:YAG laser — A free running, pulsed, 1064 nm wavelength-specific ND:YAG laser will be used. A thin 300 μm laser fiber optic will be placed parallel to the root surface, allows easy access into deep periodontal pockets. The initial pass with the laser is known as Laser Troughing, and it is done with a micro-short duration pulse, with a 4.0 watt power, 150 μs duration in pulsed mode and 20Hz frequency. Ultrasonic scaler will be then used to remove calculus. The second pass is carried out with 650 μs pulse duration, 10-30 seconds for each tooth, 4.0 watt power and 20HZ frequency, to improve the ability to generate a fibrin clot. The fibrin clot is then compressed. Relieving the occlusion is the last step of the LANAP protocol.
  Other Names: LANAP using ND:YAG laser
  Arms: Laser Assisted New Attachment Procedure using ND:YAG laser
Device: Laser Assisted New Attachment Procedure using diode laser — Diode laser (Biolase) with 940 nm wavelength, a thin flexible fiber-optic cable 300 μm attached with a power average set at 0.5-1.5 watt will be used.
  The first pass "laser troughing" is done using a thin flexible fiber-optic cable 300 μm placed parallel to the root surface, attached with a power average set at 0.5-1 watt, in continuous mode. Ultrasonic scaler will be then used to remove calculus which present on the root surface. The second pass is carried out with 1-1.5 watt power in continuous mode, 10-30 seconds for each tooth, and, to improve the ability to generate a fibrin clot. The fibrin clot is then compressed in order to enhance the healing
  Other Names: LANAP using diode laser
  Arms: Laser Assisted New Attachment Procedure using diode laser
Procedure: Scaling and Root Planing using ultrasonic and curettes — Scaling and root planing (SRP) using ultrasonic device at a moderate setting and with the appropriate tips and curettes will be also used where indicated and time spent in SRP on each tooth will not be restricted.
  Arms: Scaling and Root Planing using ultrasonic and curettes

SUMMARY:
The aim of the present study is to compare the efficacy of LANAP to conventional scaling and root planing in the management of stage II periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II generalized periodontitis PPD ≥ 5 mm with attachment loss 3-4 mm with horizontal bone loss

Exclusion Criteria:

* Patients with vertical bone loss or furcation involvement.
* History of smoking more than (10 cigarettes / day).
* Patient with medical condition that contraindicate surgical procedures.
* Patients receiving antibiotics in the past three months prior to the procedure.
* Pregnant or lactating females.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Microbiological assessment of Fusobacterium nucleatum | up to 6 months
  Subgingival plaque biofilm will be collected using paper cone after making a good isolation of the operated field and put into a sterile microcentrifuge tube containing phosphate buffered saline to be transferred immediately to the Microbiology laboratory for analysis of microbiome. Microcentrifuge tubes will be vortexed for 5 minutes then 200 ul of the resulting suspension will be subjected to DNA extraction using QIAamp DNA minikit. Specific PCR primers targeting gingival plaque associated oral microbiota (Fusobacterium nucleatum) will be used in SYBR Green Real-Time PCR. Amplification of 16SrRNA gene will be used as the denominator against which the amplification of other bacteria will be estimated. The bacterial relative quantification will be calculated automatically by the Rotor-Gene software and expressed as relative fold difference.
Microbiological assessment of Porphyromonas gingivalis | up to 6 months
  Subgingival plaque biofilm will be collected using paper cone after making a good isolation of the operated field and put into a sterile microcentrifuge tube containing phosphate buffered saline to be transferred immediately to the Microbiology laboratory for analysis of microbiome. Microcentrifuge tubes will be vortexed for 5 minutes then 200 ul of the resulting suspension will be subjected to DNA extraction using QIAamp DNA minikit. Specific PCR primers targeting gingival plaque associated oral microbiota (Porphyromonas gingivalis) will be used in SYBR Green Real-Time PCR. Amplification of 16SrRNA gene will be used as the denominator against which the amplification of other bacteria will be estimated. The bacterial relative quantification will be calculated automatically by the Rotor-Gene software and expressed as relative fold difference.
Microbiological assessment of Tannerella forsythia | up to 6 months
  Subgingival plaque biofilm will be collected using paper cone after making a good isolation of the operated field and put into a sterile microcentrifuge tube containing phosphate buffered saline to be transferred immediately to the Microbiology laboratory for analysis of microbiome. Microcentrifuge tubes will be vortexed for 5 minutes then 200 ul of the resulting suspension will be subjected to DNA extraction using QIAamp DNA minikit. Specific PCR primers targeting gingival plaque associated oral microbiota (Tannerella forsythia) will be used in SYBR Green Real-Time PCR. Amplification of 16SrRNA gene will be used as the denominator against which the amplification of other bacteria will be estimated. The bacterial relative quantification will be calculated automatically by the Rotor-Gene software and expressed as relative fold difference.

SECONDARY OUTCOMES:
Gingival index | up to 6 months
  This is used to assess the degree of gingival inflammation. Each tooth is examined and scored (0-3), where 0 = normal gingiva; 1 = mild inflammation: slight change in color, slight edema, no bleeding on probing; 2 = moderate inflammation: redness, edema, and glazing, or bleeding on probing; 3 = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding and ulceration
Plaque index | up to 6 months
  This is used to assess the amount of plaque accumulation. Each tooth is examined and scored (0-3), where 0= no plaque, 1= a thin plaque film at the free gingival margin (only seen by running a probe in the sulcus, 2= moderate plaque accumulation, 3= abundance of plaque
Clinical attachment loss | up to 6 months
  This is assessed using a Williams probe from a fixed reference point on the crown to the base of the pocket. Pocket severity is classified by the extent of clinical attachment loss in millimeters (0= normal, 1 or 2 mm = slight, 3 or 4 mm = moderate, ≥ 5 mm = severe).
Probing depth | up to 6 months
  This is measured from the margin of the gingiva to the base of the pocket using a Williams probe. The normal probing sulcus depth is considered to range from 1 to 3 mm in healthy gingiva.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt